CLINICAL TRIAL: NCT00001063
Title: A Phase II Randomized Study of the Virologic and Immunologic Effects of d4T vs Zidovudine Plus d4T vs Zidovudine Plus Ddl in HIV-Infected Patients With CD4 Cell Counts Between 300-600/mm3 and Greater Than 12 Weeks Zidovudine Experience
Brief Title: The Effectiveness of Three Drug Combinations in HIV-Infected Patients Who Have Taken Zidovudine for More Than 12 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 290; 11266 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; Stavudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the effect of stavudine (d4T) alone or with zidovudine (AZT) versus didanosine (ddI) alone or with AZT on CD4 counts, HIV RNA levels, and viral load in HIV-infected patients [AS PER AMENDMENT 3/21/97: To compare the effects of d4T alone versus ddI alone versus AZT plus ddI]. To compare the safety of d4T/AZT. AS PER AMENDMENT 3/21/97: To evaluate the pharmacokinetic interactions of AZT and d4T both at an extracellular and intracellular level.

Although AZT and ddI can delay the advancement of HIV disease, the benefit of either of these drugs has proven to be only temporary. d4T, a new nucleoside analog with a favorable toxicity profile and demonstrated activity against HIV, offers an additional therapeutic option. It is reasonably assumed that the benefit of an antiretroviral agent in terms of delaying clinical disease progression is directly related to its ability to achieve and sustain viral suppression; thus, this study measures effects on viral load and CD4 count.

DETAILED DESCRIPTION:
Although AZT and ddI can delay the advancement of HIV disease, the benefit of either of these drugs has proven to be only temporary. d4T, a new nucleoside analog with a favorable toxicity profile and demonstrated activity against HIV, offers an additional therapeutic option. It is reasonably assumed that the benefit of an antiretroviral agent in terms of delaying clinical disease progression is directly related to its ability to achieve and sustain viral suppression; thus, this study measures effects on viral load and CD4 count.

Patients are randomized in a blinded fashion to receive AZT or placebo in combination with open-label d4T or ddI for up to 48 weeks. AS PER AMENDMENT 3/21/97: The study is now composed of three arms: open-label d4T versus open-label ddI plus blinded AZT placebo versus blinded AZT plus open-label ddI. Patients originally assigned to the d4T + AZT arm, which was closed 10/96, will be given the option of discontinuing AZT and remaining on d4T monotherapy or discontinuing all study drugs. In addition, all study participants will be asked to participate in a pharmacology substudy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required for patients whose CD4 count falls below 200 cells/mm3:

* PCP prophylaxis with TMP/SMX, aerosolized pentamidine, or dapsone.

Allowed:

* Atovaquone, IV pentamidine, trimethoprim-dapsone, clindamycin-primaquine, trimetrexate, or TMP/SMX for acute PCP.
* Topical antifungals, clotrimazole, ketoconazole, fluconazole, and amphotericin B for mucosal and esophageal candidiasis.
* Itraconazole.
* Amphotericin B.
* Rifabutin.
* Isoniazid.
* Pyrazinamide.
* Clofazimine.
* Clarithromycin.
* Azithromycin.
* Ethambutol.
* Amikacin.
* Ciprofloxacin.
* Ofloxacin.
* Pyrimethamine.
* Sulfadiazine.
* Clindamycin.
* Ganciclovir.
* G-CSF.
* Acyclovir (up to 1000 mg/day).
* Erythropoietin.
* Antibiotics for bacterial infections.
* Antipyretics.
* Analgesics.
* Antiemetics.
* Rifampin.

Concurrent Treatment:

Allowed:

* Local radiation therapy.

Patients must have:

* HIV infection.
* CD4 count 300-600 cells/mm3.
* More than 12 weeks (was 24 weeks, AMENDED 3/31/96) of total prior AZT ( > 500 mg/day without serious adverse event). Subjects must be actively taking ZDV for at least 4 continuous weeks up to the time of study entry.
* No prior or current history of AIDS.
* No active opportunistic infection.
* Life expectancy of at least 2 years.
* Consent of patient and parent or guardian if less than 18 years of age.

NOTE:

* Protocol is approved for prisoner enrollment.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy requiring systemic cytotoxic chemotherapy.
* Serious underlying medical condition other than HIV that would reduce life expectancy to < 2 years.

Concurrent Medication:

Excluded:

* Antiretrovirals other than study drugs.
* Foscarnet.

Patients with the following prior conditions are excluded:

* Unexplained temperature >= 38.5 C for 7 days or chronic diarrhea (>= three stools daily) for 15 days, if occurring within 30 days prior to study entry.
* History of acute or chronic pancreatitis.
* History of grade 2 or higher peripheral neuropathy.
* History of grade 3 or worse intolerance to 500-600 mg/day AZT.

Prior Medication:

Excluded:

(within 30 days prior to study entry)

* Prior ddI, ddC, 3TC or d4T (more than 2 weeks total).
* Non-nucleoside reverse transcriptase inhibitor or protease inhibitor.
* Biologic response modifiers such as interferon and IL-2.
* Other experimental therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Study Completion 1997-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Havlir D, Study Chair; Richman D, Study Chair; Pollard R, Study Chair; Friedland G, Study Chair
Locations (33):
- United States (31):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Puerto Rico-AIDS CRS, San Juan

REFERENCES:
- [Background] d4T+AZT--unexpected CD4 drop seen in study. AIDS Treat News. 1996 Dec 20;(No 261):1. PMID 11364024
- [Background] Shaefer M, Hardy WD, Shaker-Irwin L, Williams V, Maude C, Thommes J, Graham N. HIV viral load response in subjects switched from zidovudine (ZDV)-containing to stavudine (D4T)-containing regimens in the Pacific Oaks Population Study (POPS). Int Conf AIDS. 1998;12:57 (abstract no 12228)
- [Background] Havlir DV, Friedland G, Pollard R, Tierney C, Smeaton L, Fox L, Richman DD. Combination zidovudine (ZDV) and stavudine (d4T) therapy versus other nucleosides: report of two randomized trials (ACTG 290 and 298). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:79 (abstract no 2)
- [Background] Cadman J. 2, 4, 6, 8, who's afraid to phosphorylate? GMHC Treat Issues. 1998 Feb;12(2):6-8. PMID 11365218
- [Background] Havlir DV, Tierney C, Friedland GH, Pollard RB, Smeaton L, Sommadossi JP, Fox L, Kessler H, Fife KH, Richman DD. In vivo antagonism with zidovudine plus stavudine combination therapy. J Infect Dis. 2000 Jul;182(1):321-5. doi: 10.1086/315683. Epub 2000 Jul 6. PMID 10882616
- [Background] Sommadossi JP, Zhou XJ, Moore J, Havlir DV, Friedland G, Tierney C, Smeaton L, Fox L, Richman D, Pollard R. Impairment of stavudine (d4T) phosphorylation in patients receiving a combination of zidovudine (ZDV) and d4T (ACTG 290). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:79 (abstract no 3)